CLINICAL TRIAL: NCT03881826
Title: Investigation of the Gut Microbiota in Patients With Acute Myeloid Leukemia
Acronym: MicroAML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: European Society for Clinical Nutrition and Metabolism (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B403201317128
Record Dates: First submitted 2019-02-05; First posted 2019-03-20 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Acute Myeloid Leukemia; Cachexia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haematological patients (Experimental)
  Interventions: Other: collection of clinical data and biological samples
- Healthy volunteers (Active Comparator)
  Interventions: Other: collection of clinical data and biological samples

INTERVENTIONS:
Other: collection of clinical data and biological samples — * nutritional assessement
  * cachexia symptoms
  * urine, feces and blood samples

SUMMARY:
This cohort study aims to investigate the composition and activity of the gut microbiota of patients newly diagnosed for acute myeloid leukemia (AML), in relationship with their food habits and cachectic hallmarks. The recruitment for this study is currently ongoing with the help of clinicians, nurses and data managers at the Saint-Luc clinics, University Hospital Leuven (Campus Gasthuisberg) and University Hospital Gent.

Primary Objective

•To assess the composition and activity of the gut microbiota in patients with acute myeloid leukemia (AML) compared to matched control subjects.

Secondary Objectives

* To investigate correlations between the gut microbiota, cachectic hallmarks and gut microbiota-related markers in the blood (gut permeability markers, microbial compounds, microbial metabolites).
* To characterize the changes in the gut microbial ecosystem that are induced by chemotherapy and associated with colitis.
* To assess whether the composition of the gut microbiota can predict the severity of chemotherapy-related colitis.

Study Design

This is an academic multi-centric prospective study. The study is composed of two cohorts (Fig. 1). In Cohort A, patients are included before any chemotherapy. Biological samples (urine, feces, blood) are collected, alongside information on nutritional habits, appetite and medical records. Muscle strength and body composition are also measured. Only patients receiving a standard chemotherapy are included in Cohort B. In Cohort B, biological samples are collected and body composition, muscle strength and appetite are evaluated at 2 different time points, at the end of the chemotherapy (T1) and at discharge (T4).

ELIGIBILITY:
Inclusion Criteria:

* Patients with

  * A diagnosis of AML and related precursor neoplasms according to WHO 2008 classification (excluding acute promyelocytic leukemia) including secondary AML (after an antecedent hematological disease (e.g. MDS) and therapy-related AML)
  * Acute leukemia's of ambiguous lineage according to WHO 2008
  * A diagnosis of refractory anemia with excess of blasts (MDS REAB) 2 and IPSS (International Prognostic Scoring System)-R score > 2.
* World Health Organization performance status 0, 1 or 2
* Sampled bone marrow and/ blood cells at diagnosis with molecular analysis.
* Written informed consent
* Good command of the French or Dutch language

Exclusion Criteria:

* Age < 18 years
* Age > 75 years
* Pregnancy
* Antibiotics consumption during the last 30 days before inclusion
* Recent chemotherapy (< 3 months), with exclusion of hydroxyurea
* BMI >30
* Any history of chronic intestinal affections (Crohn disease, inflammatory bowel disease, gluten intolerance)
* Gastric bypass
* Current treatment with antidiabetic or hypoglycemic drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2020-01-11 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Description of gut microbiota composition in patients with acute myeloid leukemia and control subjects | Day 0 i.e.: feces sampling is done at time of diagnosis before any chemotherapy
  Sequencing DNA extracts from patients' feces (both patients with acute myeloid leukemia and control subjects matched for BMI, sex and age) to obtain the description of gut microbiota composition in those patients
Measure of metabolites production by the gut microbiota in patients with acute myeloid leukemia and control subjects | Day 0 i.e.: feces sampling is done at time of diagnosis before any chemotherapy
  1H-NMR metabolomics performed on patients' feces (both patients with acute myeloid leukemia and control subjects matched for BMI, sex and age) to report the metabolites produced by the gut microbiota of those patients

SECONDARY OUTCOMES:
Changes in muscle strength | at day 0 (i.e.: feces sampling is done at time of diagnosis before any chemotherapy);
  Measure of muscle strength with Jamar dynamometer (in kg)
Changes in body composition | at day 0 (i.e.: feces sampling is done at time of diagnosis before any chemotherapy);
  Measure of body composition by bio-electric impedance (in kg)
Changes in appetite | at day 0 (i.e.: feces sampling is done at time of diagnosis before any chemotherapy);
  Measure of appetite with the SNAQ questionnaire (score from 5 to 20)
Changes in gut microbiota-related markers in the blood (gut permeability markers and microbial compounds) | at day 0 (i.e.: feces sampling is done at time of diagnosis before any chemotherapy);
  ELISA (in pg/ml)
Changes in gut microbiota-related markers in the blood (microbial metabolites) | at day 0 (i.e.: feces sampling is done at time of diagnosis before any chemotherapy);
  1H-NMR metabolomics
Changes in gut microbiota-related markers in urine (gut permeability markers, microbial compounds, microbial metabolites) | at day 0 (i.e.: feces sampling is done at time of diagnosis before any chemotherapy);
  ELISA and 1H-NMR metabolomics
Changes in gut microbiota composition in patients with acute myeloid leukemia before, during and after chemotherapy | at day 0 (i.e.: feces sampling is done at time of diagnosis before any chemotherapy);
  Sequencing DNA extracts from patients' feces to obtain the description of gut microbiota composition in those patients.
Changes in metabolites production by the gut microbiota in patients with acute myeloid leukemia before, during and after chemotherapy. | at day 0 (i.e.: feces sampling is done at time of diagnosis before any chemotherapy);
  1H-NMR metabolomics performed on patients' feces to report the metabolites produced by the gut microbiota of those patients.
Changes in number of participants with treatment related-related adverse events as assessed by CTCAE v4.0 | at day 0 (i.e.: feces sampling is done at time of diagnosis before any chemotherapy);
  CTCAE (common terminology criteria for adverse event version 4)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Potgens SA, Lecop S, Havelange V, Li F, Neyrinck AM, Neveux N, Maertens J, Walter J, Schoemans H, Delzenne NM, Bindels LB. Gut microbiota alterations induced by intensive chemotherapy in acute myeloid leukaemia patients are associated with gut barrier dysfunction and body weight loss. Clin Nutr. 2023 Nov;42(11):2214-2228. doi: 10.1016/j.clnu.2023.09.021. Epub 2023 Sep 25. PMID 37806074